CLINICAL TRIAL: NCT01049022
Title: Safety, Tolerability and Pharmacokinetics of Single Dose Intravenous Moxifloxacin in Pediatric Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11826; 2012-000737-40 (EudraCT Number)
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Infections
Keywords: Pharmacokinetics
MeSH Terms: conditions — Infections | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moxifloxacin (Avelox, BAY12-8039), Cohort 1 (Experimental)
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)
- Moxifloxacin (Avelox, BAY12-8039), Cohort 2 (Experimental)
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)
- Moxifloxacin (Avelox, BAY12-8039), Cohort 3 (Experimental)
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Single intravenous (IV) infusion of moxifloxacin administered over 60 minutes, at an initial dosage of 5 milligram per kilogram per body weight (mg/kg/BW) with dose escalation to 6 mg/kg in subjects of age 6 years (yrs) to less than or equal to (<=) 14 years.
  Arms: Moxifloxacin (Avelox, BAY12-8039), Cohort 1
Drug: Moxifloxacin (Avelox, BAY12-8039) — Single IV infusion of moxifloxacin administered over 60 minutes, at a dosage of 7 mg/kg/BW with dose escalation to 8 mg/kg in subjects of age 2 years to less than (<) 6 years; dose escalation was based on evaluations of the pharmacokinetic (PK) and safety data from the subjects in a preceding cohort.
  Arms: Moxifloxacin (Avelox, BAY12-8039), Cohort 2
Drug: Moxifloxacin (Avelox, BAY12-8039) — Single IV infusion of moxifloxacin administered over 60 minutes, at a dosage of 9 mg/kg/BW with dose escalation to 10 mg/kg in subjects of age 3 months to < 2 years; dose escalation was based on evaluations of the PK and safety data from the subjects in a preceding cohort.
  Arms: Moxifloxacin (Avelox, BAY12-8039), Cohort 3

SUMMARY:
The purpose of this study is to describe the pharmacokinetics of moxifloxacin in children to see what the best dose should be for children in the future. Pharmacokinetics is to see how the body absorbs, distributes, breaks down and gets rid of the study drug. The pharmacokinetics of certain drugs may be altered in children due to developmental differences in various organ functions responsible for drug elimination, as well as in general distribution characteristics. The safety of moxifloxacin in children with infections will also be looked at. Results from this study will be used to guide dosing strategies of the larger clinical trial planned for children

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ages 3 months through 14 years inclusive
* Receiving antibiotics for suspected or proven infection

Exclusion Criteria:

* Body weight greater than 45 kg
* Patients taking anti-seizure medications within 30 days of moxifloxacin dosing
* Known or suspected allergy to quinolones
* History of tendon disease/disorder related to quinolone treatment
* Severe, life-threatening disease with a life expectancy of less than 48 hours and/or known rapidly fatal underlying disease (death expected within 2 months)
* Abnormal musculoskeletal evaluation at baseline assessment; or chronic musculoskeletal disease (eg, juvenile rheumatoid arthritis); or chronic illness with high risk for chronic or recurrent arthritis or tendinitis (eg, cystic fibrosis, chronic inflammatory bowel disease)
* Cardiac arrhythmia
* Evidence of renal or hepatic disease, based on laboratory findings (serum creatinine, total bilirubin, or ALT, > 1.5 times upper limit of normal) and physical exam
* Patients receiving Class IA (e.g., quinidine, procainamide) or Class III (e.g., amiodarone, sotalol) antiarrhythmic agents
* Patients taking any medication known to increase the QT interval, eg, amiodarone, astemizole, bepridil, chloroquine, chlorpromazine, cisapride, disopyuramide, dofetilide, droperidol, halofantrine, haloperidol, ibutilide, levomethadyl, mesoradazine, methadone, pimozide, procainamide, quinidine, sotalol, terfenadine
* Pregnancy
* Clinically relevant findings in the ECG
* Participation in another clinical study during the preceding 30 days1 (last treatment from previous study to first treatment of new study)
* Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the patient's safety
* Patients taking another fluoroquinolone at the time of planned moxifloxacin dosing

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area under the Concentration-Time Curve (AUC) of Moxifloxacin and its Metabolites | Pre-dose, 1 hour (end of infusion), 1.5, 4, 8, 12 and 24 hours (Day 2) after start of infusion (samples at 36 h and 48 h were optional)
  The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Maximum Observed Drug Concentration in Plasma (Cmax) of Moxifloxacin and its Metabolites | Pre-dose, 1 hour (end of infusion), 1.5, 4, 8, 12 and 24 hours (Day 2) after start of infusion (samples at 36 h and 48 h were optional)
  Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Number of Subjects With Treatment Emergent Findings on Joint Assessment: Baseline | Baseline
  Joint assessment included formal physical examination of all joints with special care and attention to the weight-bearing joints (such as, knees, hips, and ankles) and to the shoulder girdle. All joints were examined for pain/tenderness, evidence of inflammation (i.e., redness, warmth, deformity, swelling or ballotable fluid), loss of function (to the extent this could be assessed in younger children and infants), and any restrictions to expected active/passive range of motion. An incidence count was reported as the number of subjects with at least one finding at baseline, regardless of side.
Number of Subjects With Treatment Emergent Findings on Joint Assessment : At any Time During Treatment | Day 1 up to Year 5 (follow-up)
  Joint assessment included formal physical examination of all joints with special care and attention to the weight-bearing joints (such as, knees, hips, and ankles) and to the shoulder girdle. An incidence count was reported as the number of subjects with at least one finding at any time during treatment, regardless of side.

SECONDARY OUTCOMES:
Time to Reach Maximum Drug Concentration in Plasma (tmax) of Moxifloxacin and its Metabolites | Pre-dose, 1 hour (end of infusion), 1.5, 4, 8, 12 and 24 hours (Day 2) after start of infusion (samples at 36 h and 48 h were optional)
  tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Half Life Associated With Terminal Slope (t1/2) of Moxifloxacin and its Metabolites | Pre-dose, 1 hour (end of infusion), 1.5, 4, 8, 12 and 24 hours (Day 2) after start of infusion (samples at 36 h and 48 h were optional)
  Half life associated with terminal slope refers to the elimination of the drug. It is the time taken for the blood plasma concentration to reach half the concentration in the terminal phase of elimination. It is expressed in hours (h) and derived from the terminal slope of the concentration versus time curve.
Total Amount Excreted in the Urine (Aeur) of Moxifloxacin and its Metabolites | Baseline up to 36 hour post-infusion
  Aeur refers to the total amount of moxifloxacin excreted in urine.
Volume of Distribution at Steady State (Vss) of Moxifloxacin and its Metabolites | Pre-dose, 1 hour (end of infusion), 1.5, 4, 8, 12 and 24 hours (Day 2) after start of infusion (samples at 36 h and 48 h were optional)
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the apparent volume of distribution at steady-state.
Plasma Clearance (CL) of Moxifloxacin and its Metabolites | Pre-dose, 1 hour (end of infusion), 1.5, 4, 8, 12 and 24 hours (Day 2) after start of infusion (samples at 36 h and 48 h were optional)
  Total body clearance of drug in plasma is expressed in litres per hour.
Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity Divided by Dose Per kilogram Body Weight (AUCnorm) of Moxifloxacin and its Metabolites | Pre-dose, 1 hour (end of infusion), 1.5, 4, 8, 12 and 24 hours (Day 2) after start of infusion (samples at 36 h and 48 h were optional)
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. AUCnorm is defined as AUC divided by dose per kg body weight.
Maximum Observed Plasma Concentration Divided by Dose Per kilogram Body Weight (Cmax,Norm) of Moxifloxacin and its Metabolites | Pre-dose, 1 hour (end of infusion), 1.5, 4, 8, 12 and 24 hours (Day 2) after start of infusion (samples at 36 h and 48 h were optional)
  Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Cmax,norm is defined as Cmax divided by dose (mg) per kg body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- United States (11):
  - Little Rock, Arkansas
  - Orange, California
  - San Diego, California
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Kansas City, Missouri
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Wirth S, Emil SGS, Engelis A, Digtyar V, Criollo M, DiCasoli C, Stass H, Willmann S, Nkulikiyinka R, Grossmann U; MOXIPEDIA Study Group. Moxifloxacin in Pediatric Patients With Complicated Intra-abdominal Infections: Results of the MOXIPEDIA Randomized Controlled Study. Pediatr Infect Dis J. 2018 Aug;37(8):e207-e213. doi: 10.1097/INF.0000000000001910. PMID 29356761
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/